CLINICAL TRIAL: NCT01395303
Title: Polymorphisms in the Vitamin D System and Health
Status: Completed | Type: Observational
Sponsor: University of Tromso (Other)
Responsible Party: Principal Investigator, Rolf Jorde, Professor, University of Tromso
Other Study IDs: UIT-ENDO-2011-2
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Infarction; Stroke; Diabetes; Fracture; Aortic Stenosis; Cancer; Death
Keywords: infarction; stroke; diabetes; fracture; aortic stenosis; cancer; death; vitamin D; androgens; thyroid hormones
MeSH Terms: conditions — Infarction; Stroke; Diabetes Mellitus; Fractures, Bone; Aortic Valve Stenosis; Neoplasms; Death

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA from blood clots
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- myocardial infarction: subjects with myocardial infarction in the Tromsø study end point registry
- type 2 diabetes: subjects with type 2 diabetes in the Tromsø study end point registry
- stroke: subjects with stroke in the Tromsø study end point registry
- fracture: subjects with fracture in the Tromsø study end point registry
- cancer: subjects with cancer in the Tromsø study end point registry
- death: subjects registered as dead in the Tromsø study end point registry
- aortic stenosis: subjects with aortic stenosis in the Tromsø study end point registry
- control group: randomly selected controls from the Tromsø study

SUMMARY:
Polymorphisms in the vitamin D system appear to affect the serum 25(OH)D levels. If so one would expect these polymorphisms to be associated with vitamin D related conditions and diseases, which will be tested in the present study including DNA analyses in 9700 subjects

DETAILED DESCRIPTION:
Vitamin D, which is essential in calcium metabolism, is produced in the skin after sun exposure or obtained from food, mainly fatty fish or vitamin D supplements. For activation vitamin D must be hydroxylated in the liver to 25(OH)D and thereafter in the kidney to 1,25(OH)2D. In the circulation 25(OH)D and 1,25(OH)2D are bound to a carrier protein (DBP), and for 1,25(OH)2D to exert its effect it has to bind to the vitamin D receptor (VDR).

The serum level of 25(OH)D, which is the metabolite used to evaluate a person's vitamin D status, is in part genetically determined and several polymorphisms with effects on serum 25(OH)D have been identified. These polymorphisms, where the minor allele frequencies vary between 16 and 40 %, appear as important for the serum 25(OH)D level as the effect of season, physical activity or vitamin D supplementation.

Vitamin D is not only vital for the skeleton, but appears to be related to a number of health outcomes, including mortality as previously demonstrated in the Tromsø study. However, as the serum level of 25(OH)D is strongly influenced by life-style factors that are also related to health outcomes, it is difficult to decide whether the relation between vitamin D and health is causal or not.

On the other hand, the polymorphisms are not influenced by life-style, and the effect of the polymorphisms will be life-long. Accordingly, they may be a better marker of vitamin D status than a single serum 25(OH)D measurement. Furthermore, there are a number of polymorphisms regarding the vitamin D receptor (VDR) that may be associated with health.

In the present study we will therefore relate the polymorphisms affecting the serum 25(OH)D level and the function of the VDR, with anthropometric and biochemical measures, mortality, diseases and risk factors for disease. DNA will be obtained from the 4th Tromsø study.

If we find the expected associations between the polymorphisms and diseases, this will further strengthen the role of vitamin D in human health, and may be important for recommendations regarding vitamin D supplementation. Considering the high prevalence of vitamin D deficiency world wide, this may potentially have huge consequences for public health.

The main purpose of the present study is the vitamin D system, but in the Tromsø study we have previously also found a number of associations between thyroid and androgen function and health. Obtaining DNA for analysis will be the major cost in the project, whereas analyses of individual polymorphisms are relatively cheap. We will therefore also include polymorphisms regarding thyroid and androgen function.

ELIGIBILITY:
Inclusion Criteria:

* participated in the fourth Tromsø study, later registered in our end point registry or selected as a control subject

Exclusion Criteria:

* lacking DNA sample

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects from the fourth Tromsø study performed in 1994-1995 who had blood samples taken for later DNA analyses
Sampling Method: Probability Sample
Enrollment: 9700 (Actual)
Dates: Start 2011-04; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Jorde, Professor, Principal Investigator — University of Tromso
Locations (1):
- University of Tromsø, Tromsø, Tromsø, Norway

REFERENCES:
- [Derived] Jorde R, Schirmer H, Wilsgaard T, Joakimsen RM, Mathiesen EB, Njolstad I, Lochen ML, Figenschau Y, Berg JP, Svartberg J, Grimnes G. Polymorphisms related to the serum 25-hydroxyvitamin D level and risk of myocardial infarction, diabetes, cancer and mortality. The Tromso Study. PLoS One. 2012;7(5):e37295. doi: 10.1371/journal.pone.0037295. Epub 2012 May 23. PMID 22649517